CLINICAL TRIAL: NCT07198256
Title: Research on AI-assisted Diagnosis of Common Malignant Brain Tumors Based on Magnetic Resonance Imaging
Brief Title: AI-assisted Diagnosis of Malignant Brain Tumors
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-1050
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Gliomas; Brain Metastases, Adult; Lymphoma; Brain Tumor Adult
Keywords: brain tumor; glioma; brain metastases; lymphoma; magnetic resonance imaging; artificial intelligence
MeSH Terms: conditions — Glioma; Brain Neoplasms; Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- malignant brain tumors: Retrospectively collected cases of malignant brain tumors (including gliomas, brain metastases, and brain lymphomas) that were confirmed by histopathology and had preoperative multimodal MRI images (mainly including CE-T1WI and T2-FLAIR) over the past 10 years

SUMMARY:
This study aims to establish a large-scale, multi-center MRI database for malignant brain tumors. It will develop an artificial intelligence system for the segmentation and classification of multiple subtypes of brain tumors (including glioma, metastatic tumor and lymphoma et al.) using deep learning technology. This will address the issues of small sample sizes and limited classification performance in existing methods, thereby improving the accuracy of non-invasive preoperative diagnosis, reducing the need for biopsies, and having significant clinical translational value.

DETAILED DESCRIPTION:
This study is mainly based on two centers, the Second Affiliated Hospital of Zhejiang University School of Medicine and the Zhejiang Cancer Hospital. It retrospectively collects cases of malignant brain tumors (including gliomas, brain metastases, and brain lymphomas) that have been confirmed by histopathology and have preoperative multimodal MRI images (mainly including CE-T1WI and T2-FLAIR). It is expected to include 3,000 cases. Axial CE-T1WI and T2-FLAIR images of all patients were obtained on 3.0T or 1.5T magnetic resonance imaging systems. A large-scale, multi-center MRI image database for common malignant brain tumors (gliomas, brain metastases, and brain lymphomas) was planned to be constructed. To address the automatic segmentation of complex lesion tissues in brain tumors and the auxiliary diagnosis of common malignant brain tumors, a deep learning technical approach was adopted. A deep learning-based multi-subtype brain tumor segmentation and classification diagnostic method was proposed, aiming to build an image artificial intelligence-assisted diagnostic system for common malignant brain tumors and improve the accuracy of auxiliary diagnosis of common brain malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with glioma, brain metastases, and brain lymphoma by pathology, with the patient being at least 18 years old; preoperative MRI was complete.

Exclusion Criteria:

* Poor image quality; history of previous brain surgery or radiotherapy; accompanied by other intracranial lesions.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospectively collected cases of malignant brain tumors (including gliomas, brain metastases, and brain lymphomas) that were confirmed by histopathology and had preoperative multimodal MRI images (mainly including CE-T1WI and T2-FLAIR) over the past 10 years.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Construct an AI-assisted diagnostic system for multiple subtypes of brain tumors based on deep learning. | 30 days
  Construct an AI-assisted diagnostic system for multiple subtypes of brain tumors based on deep learning, mainly including glioma, metastatic tumor and lymphoma.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang